CLINICAL TRIAL: NCT00923429
Title: A Randomized Controlled Clinical Trial of Stay-Active Care and Manual Therapy Versus Stay-Active Care Only in Subacute Low Back Pain in a Primary Health Care Setting. The Gotland Low Back Pain Study
Brief Title: Trial on Subacute Low Back Pain
Acronym: Justina
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Region Stockholm (Other Government); National Social Insurance Board, Sweden (Unknown); Uppsala County Council, Sweden (Other Government); Länsförsäkringar Research Foundation (Unknown)
Responsible Party: Kurt Svärdsudd, professor, section head, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Justina
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2009-06-18 (Estimated); Status verified 2009-06

CONDITIONS: Subacute Low Back Pain
Keywords: Manual therapy; Low back pain; Pain; Return to work
MeSH Terms: conditions — Low Back Pain; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- S-A (Active Comparator)
  Interventions: Procedure: Stay-active care
- S-A+stretch (Active Comparator)
  Interventions: Procedure: Stay-active care+stretching
- S-A+stretch+manther (Experimental)
  Interventions: Procedure: Stay-active+stretching+manual therapy
- S-A+stretch+manther+sterinject (Experimental)
  Interventions: Procedure: Stay-active+stretching+manual therapy+steroid injections

INTERVENTIONS:
Procedure: Stay-active care — No other treatment than the stay-active care
  Arms: S-A
Procedure: Stay-active care+stretching — Stay-active care and muscle stretching at home and during physiotherapist appointments
  Arms: S-A+stretch
Procedure: Stay-active+stretching+manual therapy — Manual therapy in addition to stay-active care and stretching given during GP or physiotherapist appointments and matching home exercises
  Arms: S-A+stretch+manther
Procedure: Stay-active+stretching+manual therapy+steroid injections — Manual therapy including steroid injection when indicated in addition to stay-active care and stretching during GP appointments (injections) and during GP or physiotherapist appointments (remaining treatment modalities)
  Arms: S-A+stretch+manther+sterinject

SUMMARY:
A randomized controlled trial over a 10-week period with a two-year follow-up. The objectives were to compare effects of manual therapy in addition to the stay-active concept versus the stay-active concept only in low back pain patients recruited from primary health care. 160 outpatients with acute or subacute low back pain with or without pain radiation into the legs (70 women, 90 men, ages 20-55 years) were recruited from a geographically defined area and randomly allocated to stay-active care with or without muscle stretching, or to manual therapy with or without specific corticosteroid injections in addition to the stay-active concept. Pain, disability rating index, and sickness absence measures were used as outcome at 10-week follow-up and sickness absence was measured at two-year follow-up.

DETAILED DESCRIPTION:
The study is a randomized, controlled, clinical trial in the Swedish province of Gotland, with primary data collection from 1994 to 1998. The recruitment population consisted of the 19000 employed persons born in Sweden, 20-55 years of age. Additional inclusion criteria were:

Acute or subacute perceived low back pain with or without pain radiating to one or both legs, not requiring acute surgical or rheumatological care, low back pain was required to be the dominating symptom, symptom duration of 3 months or less, preceded by at least 2 months of relative freedom from symptoms, consent to treatment and follow-up for 10 weeks, agreement not to consult other therapists during the treatment period, absence of conditions or circumstances that might jeopardize completion of treatment and follow-up, no previous treatment of current complaints with specific mobilization or manipulation, and no previous participation in the present study.

In Sweden, the National Social Insurance Offices (a government agency running the mandatory national social insurance scheme applicable to all Swedish residents) handle sick leave with a duration of two weeks or more. They as well as general practitioners (GP) and other physicians referred patients. The recruiting physician examined all patients, performed a physical examination, and made the final assessment whether they fulfilled the inclusion criteria. Of the 316 patients who were referred to the study, 111 did not meet the inclusion criteria and 45 declined participation. The 160 patients that gave informed consent were entered in the study. After baseline evaluation they were randomized by the study monitor, using sealed pre-prepared envelopes with group assignment derived from a random number table. The envelopes were inaccessible to anyone but the monitor. A design with four treatment groups was used: two experimental and two reference groups with treatment items added successively. The two-group comparison (reference vs experimental treatment) was the primary planned analysis, and pain, disability rating and sickness absence were the main outcome measures. A weighted randomization procedure was used, with 45% of the patients to reference and 55% to the experimental therapies. The Research Ethics Committee at Uppsala University approved the study.

The stay active concept was the basic management strategy in all study groups. Treatment was individual, in groups or both. Treatment modalities were chosen from a group-specific 'toolbox' after clinical assessment of the patients and according to need. Two orthopedic surgeons at Visby Hospital and eight physiotherapists treated the reference patients. In accordance with the study design, muscle stretching was a treatment option in 51% of the reference group, 41% actually received muscle stretching. Two GPs and nine physiotherapists treated the experimental patients. They received the full reference treatment, plus specific mobilization, spinal manipulation, and auto-traction when indicated. Steroid injections were a treatment option in 52% of the experimental group, 36% actually received injections.

The study population was followed over ten weeks with measurements of outcome and progression variables. Outcome measures were self-reported back pain, disability rating, return to work as assessed from sick leave records, quality of life measures, and pain drawings. Moreover, sick leave data during two years of follow up from baseline were obtained.

ELIGIBILITY:
Inclusion Criteria:

* acute or subacute perceived low back pain with or without pain radiating to one or both legs
* symptom duration of three months or less preceded by at least two months of relative freedom from symptoms
* consent to treatment and follow up for ten weeks
* agreement not to consult therapists other than those participating in the study during the treatment period

Exclusion Criteria:

* other conditions or circumstances that might jeopardize completion of treatment and follow up, such as pregnancy, malignant tumors, etcetera
* need for acute surgical or rheumatologic care
* previous treatment of current complaints with specific mobilisation or manipulation
* previous participation in the present study

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 1994-01; Primary Completion 1998-12 (Actual); Study Completion 2000-12 (Actual)

PRIMARY OUTCOMES:
Sick leave | 2 years

SECONDARY OUTCOMES:
Disability | 10 weeks
Pain | 10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Public Health and Caring Sciences, Family Medicin and Clinical Epidemiology Section, Uppsala, Sweden

REFERENCES:
- [Result] Grunnesjo MI, Bogefeldt JP, Svardsudd KF, Blomberg SI. A randomized controlled clinical trial of stay-active care versus manual therapy in addition to stay-active care: functional variables and pain. J Manipulative Physiol Ther. 2004 Sep;27(7):431-41. doi: 10.1016/j.jmpt.2004.06.001. PMID 15389174
- [Result] Grunnesjo M, Bogefeldt J, Blomberg S, Delaney H, Svardsudd K. The course of pain drawings during a 10-week treatment period in patients with acute and sub-acute low back pain. BMC Musculoskelet Disord. 2006 Aug 11;7:65. doi: 10.1186/1471-2474-7-65. PMID 16901354
- [Result] Bogefeldt J, Grunnesjo M, Svardsudd K, Blomberg S. Diagnostic differences between general practitioners and orthopaedic surgeons in low back pain patients. Ups J Med Sci. 2007;112(2):199-212. doi: 10.3109/2000-1967-194. PMID 17578820
- [Result] Bogefeldt J, Grunnesjo MI, Svardsudd K, Blomberg S. Sick leave reductions from a comprehensive manual therapy programme for low back pain: the Gotland Low Back Pain Study. Clin Rehabil. 2008 Jun;22(6):529-41. doi: 10.1177/0269215507087294. PMID 18511533
- [Derived] Grunnesjo MI, Bogefeldt JP, Blomberg SI, Strender LE, Svardsudd KF. A randomized controlled trial of the effects of muscle stretching, manual therapy and steroid injections in addition to 'stay active' care on health-related quality of life in acute or subacute low back pain. Clin Rehabil. 2011 Nov;25(11):999-1010. doi: 10.1177/0269215511403512. Epub 2011 Aug 10. PMID 21831926
- See also: Department of Public Health and Caring Sciences — http://www.pubcare.uu.se